CLINICAL TRIAL: NCT00475293
Title: A Phase 2 Clinical Trial of Panitumumab in Combination With Irinotecan Chemotherapy as 2nd-line Therapy in Subjects With Metastatic Colorectal Cancer
Brief Title: Panitumumab in Combination With Irinotecan Chemotherapy as 2nd-line Therapy in Subjects With mCRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TTD-06-04
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: metastatic colorectal cancer; 2nd-line Therapy; panitumumab; irinotecan
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Panitumumab and CPT-11

INTERVENTIONS:
Drug: Panitumumab and CPT-11 — Panitumumab will be administered by IV infusion on day 1 of each cycle just prior to the administration of chemotherapy. The starting panitumumab dose is 9 mg/kg
  Irinotecan: 350 or 300 mg/m2. day 1
  One treatment cycle is defined as the 21 day period following the commencement of treatment with panitumumab + irinotecan plus additional time, as needed, for the resolution of irinotecan-related toxicities

SUMMARY:
The purpose of this study is to assess the objective response rate (ORR) when panitumumab is administered in combination with irinotecan as 2nd-line therapy in subjects with previously treated metastatic colorectal cancer (mCRC).

DETAILED DESCRIPTION:
Aside from limited cases of resectable metastatic disease, mCRC cannot be cured with the currently available chemotherapy regimens, and there is a continued need to improve the current treatment.

Panitumumab has demonstrated objective tumour response, increase in progression free survival and has an acceptable safety profile in clinical studies in patients with metastatic colorectal cancer when used as a monotherapy or in combination with irinotecan (Meropol et al, 2003; Berlin et al, 2004; Hecht et al, 2004; Malik et al, 2005).

The addition of panitumumab to chemotherapy is expected to enhance the treatment effect of chemotherapy.

This is a Phase II, single-arm, multi-centre study. Eligible subjects will be enrolled and treated with second-line combination therapy consisting of panitumumab and irinotecan.

Prior to study entry and in order to confirm eligibility, the investigator or designee will review existing radiological images in addition to any other relevant clinical documents (reports, notes, etc.) to ensure the subject has failed or relapsed while on or after one prior chemotherapy regimen.

Panitumumab will be administered by intravenous (IV) infusion at a dose of 9 mg/kg once Q3W. Irinotecan chemotherapy (350 mg/m2) will be administered after the administration of panitumumab. Subjects will be permitted to receive panitumumab and chemotherapy until he or she develops disease progression (PD) or experiences unacceptable toxicities. Subjects who discontinue irinotecan, for example due to toxicity, will be permitted to receive panitumumab monotherapy. After discontinuation of panitumumab, the treatment period will end and subjects will attend a safety follow-up visit 56 ±3 days later.

Tumour response assessment will be performed by the investigator per the modified Response Evaluation Criteria in Solid Tumours (m-RECIST). Subjects will be evaluated for tumour response every 9 weeks ± 1 week until PD or withdrawal from the trial. Responding disease will be confirmed no less than 28 days after the criteria for response are first met. Subjects with symptoms suggestive of PD should be evaluated for tumour progression at the time the symptoms occur.

Subjects will complete an EQ-5D PRO questionnaire every 6 weeks ± 1 week, from baseline through to the end of the treatment period and at the safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman > 18 years of age
* Competent to comprehend, sign, and date an IEC-approved informed consent form
* Histologically or cytologically-confirmed metastatic adenocarcinoma of the colon or rectum.
* Radiographically documented disease progression per modified RECIST criteria either while receiving or ≤ 6 months after the last dose of prior first-line chemotherapy for mCRC
* At least 1 uni-dimensionally measurable lesion of at least 20 mm per modified RECIST criteria.
* If subject has prior history of cancer other than colorectal carcinoma, basal cell carcinoma, or cervical carcinoma in situ, then subject must not have had treatment or active disease within 5 years.
* Prior radiotherapy is acceptable.
* One and only one prior chemotherapy regimen for mCRC consisting of first-line fluoropyrimidine-based chemotherapy.
* ECOG performance status of 0, 1 or 2
* Life expectancy ≥ 3 months
* Hematologic function:ANC > 1.5 x 109/L, Platelet count > 100 x 109/L, Hemoglobin > 10 g/dL
* Renal function: Creatinine < 1.5 mg/dL
* Hepatic function: AST and ALT < 3 x ULN (if liver metastases < 5 x ULN)
* Bilirubin < 2 x ULN

Exclusion Criteria:

* No more than one prior chemotherapy regimen for mCRC consisting of first-line fluoropyrimidine-based chemotherapy. (Prior adjuvant fluoropyrimidine-based chemotherapy is allowed)
* Prior systemic therapy for the treatment of metastatic colorectal carcinoma with the exception of adjuvant fluoropyrimidine-based chemotherapy given at least 6 months prior to enrolment.
* Systemic chemotherapy, hormonal therapy, immunotherapy or experimental or approved proteins/antibodies (eg, bevacizumab) ≤ 30 days before inclusion
* Unresolved toxicities from prior systemic therapy that, in the opinion of the investigator, does not qualify the patient for inclusion
* Central nervous system/brain metastases
* Significant cardiovascular disease including unstable angina or myocardial infarction within 6 months before initiating study treatment or a history of ventricular arrhythmia
* Prior anti-EGFr antibody therapy (eg, cetuximab) or treatment small molecule EGFr tyrosine kinase inhibitors (eg, erlotinib)
* History of interstitial pneumonitis or pulmonary fibrosis or evidence of interstitial pneumonitis or pulmonary fibrosis on baseline chest CT scan
* Treatment for systemic infection within 14 days before initiating study treatment
* Radiotherapy ≤ 14 days prior to inclusion. Patients must have recovered from all radiotherapy-related toxicities
* Active inflammatory bowel disease or other bowel disease causing chronic diarrhoea (defined as > 4 loose stools per day)
* History of Gilbert's syndrome or dihydropyrimidine deficiency
* History of any medical condition that may increase the risks associated with study participation or may interfere with the interpretation of the study results
* Known positive test for human immunodeficiency virus infection, hepatitis C virus, chronic active hepatitis B infection
* subject allergic to the ingredients of the study medication or to Staphylococcus protein A
* Any co-morbid disease that would increase risk of toxicity
* Any kind of disorder that compromises the ability of the subject to give written informed consent and/or comply with the study procedures
* Any investigational agent within 30 days before enrolment
* Must not have had a major surgical procedure within 28 days of randomization
* Subject who is pregnant or breast feeding
* Woman or man of childbearing potential not consenting to use adequate contraceptive precautions i.e. double barrier contraceptive methods
* Subject unwilling or unable to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
objective response rate | 2007-2010

SECONDARY OUTCOMES:
disease control rate, duration of response, time to response, progression-free survival, time to progression,time to treatment failure,duration of stable disease | 2007-2010
adverse events | 2007-2010

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Carrato, MD, Study Chair — Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD)
Locations (1):
- Spanish Cooperative Group for Gastrointestinal Tumour Therapy, Madrid, Spain

REFERENCES:
- [Result] Carrato A, Gomez A, Escudero P, Chaves M, Rivera F, Marcuello E, Gonzalez E, Gravalos C, Constenla M, Manzano JL, Losa F, Maurel J, Duenas R, Massuti B, Gallego J, Aparicio J, Anton A, Aranda E. Panitumumab and irinotecan every 3 weeks is an active and convenient regimen for second-line treatment of patients with wild-type K-RAS metastatic colorectal cancer. Clin Transl Oncol. 2013 Sep;15(9):705-11. doi: 10.1007/s12094-012-0993-x. Epub 2013 Jan 29. PMID 23359181
- See also: Related Info — http://www.ttdgroup.org